CLINICAL TRIAL: NCT03614182
Title: Effects of Simultaneous or Sequential Combination of Physical and Cognitive Training on Dual-task Walking Performance for Community-dwelling Healthy Older Adults: a Randomized Controlled Trial.
Brief Title: Effects of Simultaneous or Sequential Combination of Physical and Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Li-Ling Chuang, Associated Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201702091B0
Record Dates: First submitted 2018-07-31; First posted 2018-08-03 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Healthy Older Adults
MeSH Terms: interventions — Cognitive Training; Precision Medicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- physical training concurrent with cognitive training (Experimental): The physical training concurrent with cognitive training group (the P+C group) will receive training at progressively increasing task difficulty 3 times a week for 12 weeks and followed by another 12 weeks without exercise (follow-up).
  Interventions: Device: physical training concurrent with cognitive training
- physical training followed by cognitive training (Active Comparator): The physical training followed by cognitive training will receive training at progressively increasing task difficulty 3 times a week for 12 weeks and followed by another 12 weeks without exercise (follow-up).
  Interventions: Device: physical training followed by cognitive training
- physical training without cognitive training (Active Comparator): The physical training without cognitive training group will receive training at progressively increasing task difficulty 3 times a week for 12 weeks and followed by another 12 weeks without exercise (follow-up).
  Interventions: Device: physical training without cognitive training

INTERVENTIONS:
Device: physical training concurrent with cognitive training — The P+C group will undertake standing balance, stepping, and treadmill walking training while concurrently perform cognitive tasks.
  Other Names: P+C
  Arms: physical training concurrent with cognitive training
Device: physical training followed by cognitive training — The P-then-C group will train the same set of standing balance, stepping, and treadmill walking activities as the P+C group while followed by cognitive training later.
  Other Names: P-then-C
  Arms: physical training followed by cognitive training
Device: physical training without cognitive training — The P group will only train the same set of standing balance, stepping, and treadmill walking activities as the other two groups.
  Other Names: P
  Arms: physical training without cognitive training

SUMMARY:
The objective of this study is to investigate psychometric properties of dual-task walking assessments and compare effects of simultaneous or sequential combination of physical and cognitive training on dual-task walking and cognitive performance for community-dwelling healthy older adults.

DETAILED DESCRIPTION:
English Synopsis

I. Title of Study:

Effects of simultaneous or sequential combination of physical and cognitive training on dual-task walking performance for community-dwelling healthy older adults: a randomized controlled trial.

II. Study Objectives:

The objective of this study is to investigate psychometric properties of dual-task walking assessments and compare effects of simultaneous or sequential combination of physical and cognitive training on dual-task walking and cognitive performance for community-dwelling healthy older adults. Specifically, the study aims to test: 1) the psychometric properties (i.e., test-retest reliability and validity) of dual-task walking outcome measures, 2) the effectiveness of delivering physical and cognitive training via simultaneous or sequential way (physical training concurrent to or followed by a cognitive training) on improving dual-task walking for healthy older adults by using good psychometric properties of outcome measures, 3) the changed CMI pattern of older adults after simultaneous or sequential physical and cognitive training.

III. Study Design A metric analysis and comparative efficacy research will be conducted at medical center(s). Sixty community-dwelling ambulatory healthy older adults will receive dual-task walking assessments twice at pretreatment with a 1-week interval for test-retest assessment and investigation of the reliability and validity of outcome measures. The primary outcome measure of the six dual-task walking assessments will include two types of walking conditions (walking at preferred speed and fast speed) and simultaneously perform three cognitive tasks (Serial Three Subtractions, Stroop, and Auditory Stroop tasks). These three cognitive tasks represent different domains of cognitive function: working memory and executive function. Concurrent validity will be studied to validate the dual-task walking measures with each other and with the item 14 of the mini-Balance Evaluation Systems test (Mini-BESTest) and dual-task Timed-up-and-Go test (dual-TUG) obtain concurrently for assessing dual-task ability. In addition, we will compare dual-task walking performance between older fallers and non-fallers to examine discriminant validity of dual-task assessments.

A comparative efficacy research is a single-blind, randomized controlled trial. Sixty healthy elderly will be randomized to physical training concurrent with cognitive training (P+C, n=20), or physical training followed by cognitive training (P-then-C, n=20), or physical training without cognitive training (P, n=20) groups. The P+C group will undertake standing balance, stepping, and treadmill walking training while concurrently perform cognitive tasks. The P-then-C group will train the same set of standing balance, stepping, and treadmill walking activities as the P+C group while followed by cognitive training later. The P group will only train the same set of standing balance, stepping, and treadmill walking activities as the other two groups. All three groups will receive training at progressively increasing task difficulty 3 times a week for 12 weeks and followed by another 12 weeks without exercise (follow-up). Two baselines, 12 week, and 24 week data will be analyzed using multivariate statistical analyses and groups will be compared on treatment related changes in dual-task walking and cognitive performance among participants. To determine comparative effectiveness of interventions on primary outcomes (dual-task walking speed and composite score of cognitive tasks), two way mixed repeated measure ANOVAs will be used.

A blinded assessor will administer four assessments. All participants will be examined gait and cognitive performance under single-task (walking only, cognitive tasks only) and dual-task conditions (walking while performing 3 cognitive tasks) at two baselines, post intervention, and 3-month follow-up. The primary outcome measure of gait and cognition is gait speed and composite score of accuracy and reaction time of the cognitive tasks under single- and dual-task conditions. The secondary outcome measures will be the Berg Balance Scale, Mini-BESTest, dual-TUG, Functional Gait Assessment, Physical Activity Scale for the Elderly, Activities-Specific Balance Confidence Scale, Chair Stand Test, hand-held dynamometers, and Geriatric Depression Scale Short Form. Repeated measure ANOVA will be used to compare measurements at baseline, after training, and follow-up among the groups.

Number of Planned Patients: 60 healthy older adults Duration of the Study: 2018/08/01～2021/07/31

ELIGIBILITY:
Inclusion Criteria:

* age more than 65 years old
* able to walk 10 m;
* no severe vision, hearing, cognition, and language problems.

Exclusion Criteria:

* neurological or musculoskeletal diagnosis that affects walking
* unable standing for at least 2 minutes,
* MMSE score <24 or severe uncorrected visual deficits
* moderate to severe high blood pressure (systolic pressure ≧ 160mmHg and diastolic blood pressure ≧ 100mmHg )

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
gait speed | 5 minutes
  Participants will walk 10m at their preferred speed and at fast speed. A 12-meter walkway will be used for walking testing. In order to allow the subjects to have enough distance to accelerate and decelerate, only the time taken to walk the middle 10 meters will be recorded by a stopwatch. The primary gait parameter is gait speed (cm/s) under dual-task walking conditions using the 10 Meter Walking Test,
composite score | 10 minutes
  A composite score for cognitive-task performance will be calculated by dividing the accuracy (% correct responses) with the reaction time of correct answers (milliseconds), which accounts for speed-accuracy trade-offs in the overall dual-task effect.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS). | 5-10 minutes
  The BBS is a 14-item scale quantitatively assesses both static and dynamic balance. The items are scored from 0 to 4, with a score of 0 representing independent item completion. Scores of the BBS range from 0 to 56, with higher scores suggest better balance.
Mini-Balance Evaluation Systems Test (Mini-BESTest). | 10 minutes
  The Mini-BESTest consists of 14 items and includes four subscales: anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait. Each item is rated on a three-point ordinal scale (0 = severe, 1=moderate, and 2 = normal), with a maximum score of 28 points.
Timed Up and Go Test (TUG). | 2 minutes
  The TUG test will be used as an index of dynamic balance of the elderly. At the signal, participants stand up, walk 3m, turn, walk back, and sit down again. The score is the time to complete the test measured using a stopwatch. The TUG test will be administered under the single-task (preferred speed and maximum fast) and dual-task conditions (tray carrying and counting backward by 3s). In dual-task condition, participants will be asked to perform the TUG test while carrying a tray with glasses (dual-TUG manual) or counting backward by 3s (dual-TUG cognition). The instruction for dual-TUG tests is to walk with your comfortable speed and concurrently perform a secondary task (carry the tray in front of you with both hands without dropping glasses on the tray or counting backward by 3s).
Functional Gait Assessment (FGA). | 10 minutes
  The FGA is comprised of 10-item that contains 7 of 8 items (except walking around obstacles) from the Dynamic Gait Index and 3 additional tasks, including walking with a narrow base of support, walking with the eyes closed, and walking backward. Subjects' performance of each test item was rated on a 4-point scale (0-3), with the total score ranging between 0 and 30.
Physical Activity Scale for the Elderly (PASE). | 5 minutes
  The Chinese version of the PASE (PASE-C) will with good test-retest reliability and concurrent validity be used to quantify activity levels for the elderly
Chair Stand Test (CS) | 2 minutes
  The Chair Stand Test measures lower extremity muscular strength. The participants will be instructed to stand from a seated on the chair position as much as possible for 30 seconds. The total number of stands was counted in 30 seconds. Timed five-chair stand (TCS) is the time measured using a stopwatch to complete five times of standing from sitting.
Muscle Strength of Lower-Extremity | 10 minutes
  Handheld dynamometers (MicroFET2, Hoggan Health Industries Inc, West Jordan, Utah; Jamar ® Plus+ hand dynamometer, Patterson Medical® Sammons Preston®) will be used to measure the maximum isometric strength of tibialis anterior and grip Handheld dynamometers (MicroFET2, Hoggan Health Industries Inc, West Jordan, Utah; Jamar ® Plus+ hand dynamometer, Patterson Medical® Sammons Preston®) will be used to measure the maximum isometric strength of tibialis anterior and grip strength (averaged over three attempts and left and right limbs) using a standard protocol with high test-retest reliability.
Activity-specific Balance Confidence Scale (ABC). | 2 minutes
  The ABC will be used to determine fear of falling and self-reported confidence when performing 15 different daily activities, such as walking around the house, walking up and down stairs, and walking on slippery floors. A confidence rating scale ranges from 0% to 100%, with 0% indicating no confidence, and 100% indicating full confidence.
Geriatric Depression Scale Short Form (GDS-SF). | 2 minutes
  Previous studies showed that physical activity is negatively associated with mental disorder, such as depressive symptoms in older adults. Depressive symptoms will be assessed using the 15-item GDS-SF rating from 0 to 15.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No